CLINICAL TRIAL: NCT00712101
Title: Prospective Randomized Controlled Clinical Study to Compare Abciximab-bolus i.v. Versus i.c. in Primary PCI in Patients With Acute ST-elevation Myocardial Infarction
Brief Title: Abciximab i.v. Versus i.c. in ST-elevation Myocardial Infarction
Acronym: AIDA STEMI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Leipzig (Other)
Responsible Party: Dr. Holger Thiele, University of Leipzig - Heart Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Final version 1.1
Record Dates: First submitted 2008-07-03; First posted 2008-07-09 (Estimated); Last update posted 2011-04-20 (Estimated); Status verified 2009-08

CONDITIONS: ST-elevation Myocardial Infarction
Keywords: infarction; intervention; stent; abciximab; platelets
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Abciximab bolus administration intracoronary
  Interventions: Drug: abciximab intracoronary
- 2 (Active Comparator): Abciximab bolus intravenously
  Interventions: Drug: abciximab intravenously

INTERVENTIONS:
Drug: abciximab intracoronary — administer abciximab bolus intracoronary during primary percutaneous coronary intervention
  Arms: 1
Drug: abciximab intravenously — administer abciximab bolus intravenously during primary percutaneous coronary intervention
  Arms: 2

SUMMARY:
The purpose of this study is to examine whether intracoronary abciximab bolus application with subsequent 12 hour intravenous infusion in addition to primary percutaneous coronary intervention is beneficial for patients with STEMI in comparison to standard i.v. bolus application with respect to 90-day mortality, reinfarction and new congestive heart failure.

DETAILED DESCRIPTION:
In patients with acute ST-elevation myocardial infarction (STEMI) primary percutaneous coronary intervention (PCI) is the preferred reperfusion regimen, if performed by experienced operators in a timely manner. Nevertheless, myocardial damage is not immediately terminated after successful epicardial reperfusion by primary PCI. Current strategies are directed to improve myocardial tissue perfusion, which is impaired in approximately 50% of patients and which has prognostic impact. Adjunctive intravenous abciximab administration is an established therapy to improve coronary microcirculation and reduce major cardiac adverse events.5-10 In randomized clinical trials intravenous abciximab administration has been studied. Clinical trials have shown that earlier administration results in higher preinterventional TIMI-flow with subsequent improved perfusion post PCI. However, in a pooled analysis there was no effect on mortality. As door-to-balloon-times getting shorter in current trials, earlier abciximab administration requires treatment in the prehospital setting, which poses substantial logistic obstacles. Another option might be intracoronary abciximab bolus administration which results in very high local platelet inhibitor concentrations. This might be favorable in dissolution of thrombi and microemboli with subsequent improved myocardial microcirculation, reduction of no-reflow, and infarct size. Currently, there is only limited clinical experience on the efficacy of intracoronary abciximab administration mainly restricted to case reports, retrospective registries or small randomized trials. In a recently published randomized clinical trial, we were able to show that intracoronary versus intravenous abciximab bolus administration has beneficial effects on the occurrence of no-reflow and infarct size assessed by contrast-enhancement magnetic resonance imaging. This led to a trend towards improved clinical outcome. The composite major adverse cardiac event rate, defined as death, reinfarction, target vessel revascularization, and new congestive heart failure, at 30 day follow-up was 15.6% after intravenous and 5.2% after intracoronary abciximab administration (relative risk 3.00; 95% confidence intervals 0.94-10.80; p=0.06).

Currently, there is no adequately powered clinical trial to assess the effects of intracoronary bolus in comparison to standard intravenous abciximab administration. Due to its general availability and its ease of intracoronary administration this treatment has overwhelming potential in clinical practice, which is much easier to achieve than a logistically cumbersome prehospital or interhospital transfer administration.

In the era of evidence-based medicine, such a trial is of paramount importance to achieve a break-through in abciximab use and a reduction of the high associated morbidity and mortality of STEMI patients.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical symptoms:

   * Angina pectoris < 12 hours and
   * Persistent angina > 30 minutes
2. ECG-criteria for ST-elevation myocardial infarction in 12-lead ECG:

   * ST-segment elevation > 1mm in ≥ 2 extremity leads and/or
   * ST-segment elevation > 2mm in ≥ 2 adjacent precordial leads
3. Informed consent

Exclusion Criteria:

1. No informed consent
2. Pregnancy
3. Known allergy to abciximab, ASA or heparin
4. Active peptic ulcus ventriculi or duodeni
5. Active, non-superficial bleeding
6. History of major surgery (including intracranial or intraspinal) <4 weeks
7. active internal bleeding
8. Cerebrovascular complications < 2 years
9. Known coagulation defect or thrombocytopenia
10. Arteriovenous malformations or aneurysm
11. Severe liver insufficiency, renal insufficiency requiring dialysis
12. Uncontrolled hypertension, hypertensive retinopathy
13. Vaskulitis
14. Thrombolysis < 12 h
15. Participation in another trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1912 (Estimated)
Dates: Start 2008-07; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Combined clinical endpoint: death, reinfarction, new congestive heart failure | 90 days

SECONDARY OUTCOMES:
ST-segment resolution 90 minute ECG TIMI-flow post PCI indirect infarct size by enzyme release individual clinical endpoints | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Holger Thiele, MD, PhD, Study Chair — Heart Center Leipzig - University Hospital; Gerhard Schuler, MD, PhD, Study Director — Heart Center Leipzig - University Hospital; Jochen Woehrle, MD, PhD, Principal Investigator — University of Ulm
Locations (11):
- Germany (11):
  - Zentralklinik Bad Berka, Bad Berka
  - Herz- und Gefäß-KLinik Bad Neustadt, Bad Neustadt an der Saale
  - Herz und Diabeteszentrum Bad Oeynhausen, Bad Oeynhausen
  - Klinikum Links der Weser - Bremen, Bremen
  - Klinikum Coburg, Coburg
  - University of Leipzig - Heart Center, Leipzig
  - Carl-von-Basedow-Klinikum Merseburg, Merseburg
  - Klinikum Pirna, Pirna
  - Krankenhaus der Barmherzigen Brüder, Regensburg
  - Jochen Wöhrle, Ulm
  - Klinikum der Stadt Villingen-Schwenningen, Villingen-Schwenningen

REFERENCES:
- [Background] Thiele H, Schindler K, Friedenberger J, Eitel I, Furnau G, Grebe E, Erbs S, Linke A, Mobius-Winkler S, Kivelitz D, Schuler G. Intracoronary compared with intravenous bolus abciximab application in patients with ST-elevation myocardial infarction undergoing primary percutaneous coronary intervention: the randomized Leipzig immediate percutaneous coronary intervention abciximab IV versus IC in ST-elevation myocardial infarction trial. Circulation. 2008 Jul 1;118(1):49-57. doi: 10.1161/CIRCULATIONAHA.107.747642. Epub 2008 Jun 16. PMID 18559698
- [Derived] Lange T, Backhaus SJ, Schulz A, Evertz R, Kowallick JT, Bigalke B, Hasenfuss G, Thiele H, Stiermaier T, Eitel I, Schuster A. Cardiovascular magnetic resonance-derived left atrioventricular coupling index and major adverse cardiac events in patients following acute myocardial infarction. J Cardiovasc Magn Reson. 2023 Apr 13;25(1):24. doi: 10.1186/s12968-023-00929-w. PMID 37046343
- [Derived] Backhaus SJ, Rosel SF, Stiermaier T, Schmidt-Rimpler J, Evertz R, Schulz A, Lange T, Kowallick JT, Kutty S, Bigalke B, Gutberlet M, Hasenfuss G, Thiele H, Eitel I, Schuster A. Left-atrial long-axis shortening allows effective quantification of atrial function and optimized risk prediction following acute myocardial infarction. Eur Heart J Open. 2022 Aug 12;2(5):oeac053. doi: 10.1093/ehjopen/oeac053. eCollection 2022 Sep. PMID 36268539
- [Derived] Backhaus SJ, Aldehayat H, Kowallick JT, Evertz R, Lange T, Kutty S, Bigalke B, Gutberlet M, Hasenfuss G, Thiele H, Stiermaier T, Eitel I, Schuster A. Artificial intelligence fully automated myocardial strain quantification for risk stratification following acute myocardial infarction. Sci Rep. 2022 Jul 18;12(1):12220. doi: 10.1038/s41598-022-16228-w. PMID 35851282
- [Derived] Jensch PJ, Stiermaier T, Reinstadler SJ, Feistritzer HJ, Desch S, Fuernau G, de Waha-Thiele S, Thiele H, Eitel I. Prognostic relevance of peri-infarct zone measured by cardiovascular magnetic resonance in patients with ST-segment elevation myocardial infarction. Int J Cardiol. 2022 Jan 15;347:83-88. doi: 10.1016/j.ijcard.2021.11.017. Epub 2021 Nov 10. PMID 34767896
- [Derived] Lange T, Stiermaier T, Backhaus SJ, Boom PC, Kowallick JT, de Waha-Thiele S, Lotz J, Kutty S, Bigalke B, Gutberlet M, Feistritzer HJ, Desch S, Hasenfuss G, Thiele H, Eitel I, Schuster A. Functional and prognostic implications of cardiac magnetic resonance feature tracking-derived remote myocardial strain analyses in patients following acute myocardial infarction. Clin Res Cardiol. 2021 Feb;110(2):270-280. doi: 10.1007/s00392-020-01747-1. Epub 2020 Oct 20. PMID 33083869
- [Derived] Schuster A, Lange T, Backhaus SJ, Strohmeyer C, Boom PC, Matz J, Kowallick JT, Lotz J, Steinmetz M, Kutty S, Bigalke B, Gutberlet M, de Waha-Thiele S, Desch S, Hasenfuss G, Thiele H, Stiermaier T, Eitel I. Fully Automated Cardiac Assessment for Diagnostic and Prognostic Stratification Following Myocardial Infarction. J Am Heart Assoc. 2020 Sep 15;9(18):e016612. doi: 10.1161/JAHA.120.016612. Epub 2020 Sep 2. PMID 32873121
- [Derived] Backhaus SJ, Kowallick JT, Stiermaier T, Lange T, Navarra JL, Koschalka A, Evertz R, Lotz J, Kutty S, Hasenfuss G, Gutberlet M, Thiele H, Eitel I, Schuster A. Cardiac Magnetic Resonance Myocardial Feature Tracking for Optimized Risk Assessment After Acute Myocardial Infarction in Patients With Type 2 Diabetes. Diabetes. 2020 Jul;69(7):1540-1548. doi: 10.2337/db20-0001. Epub 2020 Apr 24. PMID 32335515
- [Derived] Schuster A, Backhaus SJ, Stiermaier T, Kowallick JT, Stulle A, Koschalka A, Lotz J, Kutty S, Bigalke B, Gutberlet M, Hasenfuss G, Thiele H, Eitel I. Fast manual long-axis strain assessment provides optimized cardiovascular event prediction following myocardial infarction. Eur Heart J Cardiovasc Imaging. 2019 Nov 1;20(11):1262-1270. doi: 10.1093/ehjci/jez077. PMID 31329854
- [Derived] Backhaus SJ, Kowallick JT, Stiermaier T, Lange T, Koschalka A, Navarra JL, Lotz J, Kutty S, Bigalke B, Gutberlet M, Feistritzer HJ, Hasenfuss G, Thiele H, Schuster A, Eitel I. Culprit vessel-related myocardial mechanics and prognostic implications following acute myocardial infarction. Clin Res Cardiol. 2020 Mar;109(3):339-349. doi: 10.1007/s00392-019-01514-x. Epub 2019 Jul 5. PMID 31278521
- [Derived] Reinstadler SJ, Stiermaier T, Eitel C, Fuernau G, Saad M, Poss J, de Waha S, Mende M, Desch S, Metzler B, Thiele H, Eitel I. Impact of Atrial Fibrillation During ST-Segment-Elevation Myocardial Infarction on Infarct Characteristics and Prognosis. Circ Cardiovasc Imaging. 2018 Feb;11(2):e006955. doi: 10.1161/CIRCIMAGING.117.006955. PMID 29391346
- [Derived] Stiermaier T, Jobs A, de Waha S, Fuernau G, Poss J, Desch S, Thiele H, Eitel I. Optimized Prognosis Assessment in ST-Segment-Elevation Myocardial Infarction Using a Cardiac Magnetic Resonance Imaging Risk Score. Circ Cardiovasc Imaging. 2017 Nov;10(11):e006774. doi: 10.1161/CIRCIMAGING.117.006774. PMID 29122844
- [Derived] Reinstadler SJ, Stiermaier T, Eitel C, Metzler B, de Waha S, Fuernau G, Desch S, Thiele H, Eitel I. Relationship between diabetes and ischaemic injury among patients with revascularized ST-elevation myocardial infarction. Diabetes Obes Metab. 2017 Dec;19(12):1706-1713. doi: 10.1111/dom.13002. Epub 2017 Jul 25. PMID 28474817
- [Derived] Reinstadler SJ, Stiermaier T, Eitel C, Saad M, Metzler B, de Waha S, Fuernau G, Desch S, Thiele H, Eitel I. Antecedent hypertension and myocardial injury in patients with reperfused ST-elevation myocardial infarction. J Cardiovasc Magn Reson. 2016 Nov 11;18(1):80. doi: 10.1186/s12968-016-0299-1. PMID 27832796
- [Derived] de Waha S, Eitel I, Desch S, Fuernau G, Poss J, Schuler G, Thiele H. Impact of multivessel coronary artery disease on reperfusion success in patients with ST-elevation myocardial infarction: A substudy of the AIDA STEMI trial. Eur Heart J Acute Cardiovasc Care. 2017 Oct;6(7):592-600. doi: 10.1177/2048872615624240. Epub 2015 Dec 21. PMID 26691729
- [Derived] Poss J, Desch S, Eitel C, de Waha S, Thiele H, Eitel I. Left Ventricular Thrombus Formation After ST-Segment-Elevation Myocardial Infarction: Insights From a Cardiac Magnetic Resonance Multicenter Study. Circ Cardiovasc Imaging. 2015 Oct;8(10):e003417. doi: 10.1161/CIRCIMAGING.115.003417. PMID 26481162
- [Derived] Jobs A, Eitel C, Poss J, Desch S, Thiele H, Eitel I. Effect of Pericardial Effusion Complicating ST-Elevation Myocardial Infarction as Predictor of Extensive Myocardial Damage and Prognosis. Am J Cardiol. 2015 Oct 1;116(7):1010-6. doi: 10.1016/j.amjcard.2015.07.007. Epub 2015 Jul 15. PMID 26235929
- [Derived] Eitel I, Poss J, Jobs A, Eitel C, de Waha S, Barkhausen J, Desch S, Thiele H. Left ventricular global function index assessed by cardiovascular magnetic resonance for the prediction of cardiovascular events in ST-elevation myocardial infarction. J Cardiovasc Magn Reson. 2015 Jul 16;17(1):62. doi: 10.1186/s12968-015-0161-x. PMID 26174798
- [Derived] Rommel KP, Badarnih H, Desch S, Gutberlet M, Schuler G, Thiele H, Eitel I. QRS complex distortion (Grade 3 ischaemia) as a predictor of myocardial damage assessed by cardiac magnetic resonance imaging and clinical prognosis in patients with ST-elevation myocardial infarction. Eur Heart J Cardiovasc Imaging. 2016 Feb;17(2):194-202. doi: 10.1093/ehjci/jev135. Epub 2015 Jun 9. PMID 26060202
- [Derived] Eitel I, de Waha S, Wohrle J, Fuernau G, Lurz P, Pauschinger M, Desch S, Schuler G, Thiele H. Comprehensive prognosis assessment by CMR imaging after ST-segment elevation myocardial infarction. J Am Coll Cardiol. 2014 Sep 23;64(12):1217-26. doi: 10.1016/j.jacc.2014.06.1194. PMID 25236513
- [Derived] Rommel KP, Baum A, Mende M, Desch S, Gutberlet M, Schuler G, Thiele H, Eitel I. Prognostic significance and relationship of worst lead residual ST segment elevation with myocardial damage assessed by cardiovascular MRI in myocardial infarction. Heart. 2014 Aug;100(16):1257-63. doi: 10.1136/heartjnl-2013-305462. Epub 2014 Jun 4. PMID 25049315
- [Derived] Fuernau G, Eitel I, Wohrle J, Kerber S, Lauer B, Pauschinger M, Schwab J, Birkemeyer R, Pfeiffer S, Mende M, Brosteanu O, Neuhaus P, Desch S, de Waha S, Gutberlet M, Schuler G, Thiele H. Impact of long-term statin pretreatment on myocardial damage in ST elevation myocardial infarction (from the AIDA STEMI CMR Substudy). Am J Cardiol. 2014 Aug 15;114(4):503-9. doi: 10.1016/j.amjcard.2014.05.026. Epub 2014 Jun 6. PMID 24994545
- [Derived] Eitel I, Gehmlich D, Amer O, Wohrle J, Kerber S, Lauer B, Pauschinger M, Schwab J, Birkemeyer R, Zimmermann R, Mende M, de Waha S, Desch S, Gutberlet M, Schuler G, Thiele H. Prognostic relevance of papillary muscle infarction in reperfused infarction as visualized by cardiovascular magnetic resonance. Circ Cardiovasc Imaging. 2013 Nov;6(6):890-8. doi: 10.1161/CIRCIMAGING.113.000411. Epub 2013 Aug 23. PMID 23973868
- [Derived] Eitel I, Wohrle J, Suenkel H, Meissner J, Kerber S, Lauer B, Pauschinger M, Birkemeyer R, Axthelm C, Zimmermann R, Neuhaus P, Brosteanu O, de Waha S, Desch S, Gutberlet M, Schuler G, Thiele H. Intracoronary compared with intravenous bolus abciximab application during primary percutaneous coronary intervention in ST-segment elevation myocardial infarction: cardiac magnetic resonance substudy of the AIDA STEMI trial. J Am Coll Cardiol. 2013 Apr 2;61(13):1447-54. doi: 10.1016/j.jacc.2013.01.048. Epub 2013 Feb 27. PMID 23466078
- [Derived] Thiele H, Wohrle J, Hambrecht R, Rittger H, Birkemeyer R, Lauer B, Neuhaus P, Brosteanu O, Sick P, Wiemer M, Kerber S, Kleinertz K, Eitel I, Desch S, Schuler G. Intracoronary versus intravenous bolus abciximab during primary percutaneous coronary intervention in patients with acute ST-elevation myocardial infarction: a randomised trial. Lancet. 2012 Mar 10;379(9819):923-931. doi: 10.1016/S0140-6736(11)61872-2. Epub 2012 Feb 21. PMID 22357109
- [Derived] Desch S, Siegemund A, Scholz U, Adam N, Eitel I, de Waha S, Furnau G, Lurz P, Wetzel S, Schuler G, Thiele H. Platelet inhibition and GP IIb/IIIa receptor occupancy by intracoronary versus intravenous bolus administration of abciximab in patients with ST-elevation myocardial infarction. Clin Res Cardiol. 2012 Feb;101(2):117-24. doi: 10.1007/s00392-011-0372-6. Epub 2011 Oct 21. PMID 22015616
- [Derived] Thiele H, Wohrle J, Neuhaus P, Brosteanu O, Sick P, Prondzinsky R, Birkemeyer R, Wiemer M, Kerber S, Schuehlen H, Kleinertz K, Axthelm C, Zimmermann R, Rittger H, Braun-Dullaeus RC, Lauer B, Burckhardt W, Ferrari M, Bergmann MW, Hambrecht R, Schuler G; Abciximab Intracoronary versus intravenously Drug Application in ST-Elevation Myocardial Infarction (AIDA STEMI) Investigators. Intracoronary compared with intravenous bolus abciximab application during primary percutaneous coronary intervention: design and rationale of the Abciximab Intracoronary versus intravenously Drug Application in ST-Elevation Myocardial Infarction (AIDA STEMI) trial. Am Heart J. 2010 Apr;159(4):547-54. doi: 10.1016/j.ahj.2009.12.038. PMID 20362711